CLINICAL TRIAL: NCT00974506
Title: Pilot Study Complementary Therapies in Geriatric Patients
Brief Title: Pilot Study: Complementary Therapies in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Homöopathie Stiftung (Unknown); omoeon e.V. (Unknown)
Responsible Party: Claudia M. Witt, MD, Institute for Social Medicine, Epidemiology, and Health Economics, Charité
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMGER09
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2009-09

CONDITIONS: Geriatric Patients
Keywords: geriatric patients living in residential community (shared flats), multiple disease-conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAM-intervention (Active Comparator): Complex intervention containing exercise therapy, nutritional advice, homeopathic treatment, naturopathic treatment in addition to routine therapy by general practitioner
  Interventions: Other: CAM-intervention
- Routine care therapy (Active Comparator): Routine care therapy by general practitioner
  Interventions: Other: Routine care therapy

INTERVENTIONS:
Other: CAM-intervention — Complex intervention containing exercise therapy, nutritional advice, homeopathic treatment, naturopathic treatment in addition to routine care therapy by general practitioner
  Arms: CAM-intervention
Other: Routine care therapy — Routine care therapy by general practitioner
  Arms: Routine care therapy

SUMMARY:
In a randomized controlled pilot study the investigators include geriatric patients living in a geriatric residential community. Two interventions are compared:

1. a complex intervention containing exercise therapy, nutritional advice, homeopathy and naturopathy in addition to routine therapy by the general practitioner
2. routine care by general practitioner

The investigators assess the effect of the complex intervention on activities of daily living (AMPS, Barthel Index, Nosger), quality of life (Qualidem, Profile of Wellbeing), risk of falls (Tinetti), falls, cognition (Minimental Status Test), hospital admissions, medication use.

The results of this exploratory study are needed to plan a randomized controlled trial (RCT) with confirmatory design in the future.

ELIGIBILITY:
Inclusion Criteria:

* living in shared flat/residential community
* informed consent of patient or authorized representative

Exclusion Criteria:

* participation in another study within the last 6 months
* acute or chronic disease condition that does not allow participation
* actual use of complementary therapies

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

SECONDARY OUTCOMES:
Assessment of motor and process skills (AMPS) | 3, 6, 12 months
Qualidem | 3, 6, 12 months
Barthel Index | 3, 6, 12 months
Nurses Observation Scale for Geriatric Patients | 3, 6, 12 months
Minimental Status Test | 12 months
Tinetti Test | 3, 6, 12 months
Profile of Wellbeing | 3, 6, 12 months
Medication use and Potentially Inappropriate Medication Use (Beers Criteria 2003) | 3, 6, 12 months
Falls (Esslinger Sturzprotokoll) | 12 months
hospital admissions | 12 months
Adverse effects | 12 months
Interviews with health care team and relatives. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany
Locations (1):
- Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, State of Berlin, Germany